CLINICAL TRIAL: NCT04227327
Title: A Phase 2, Open Label, Multicenter, Single Arm Trial Evaluating the Activity and Safety of Abemaciclib + Aromatase Inhibitors (AIs) After 1st-line Treatment With High-Dose Fulvestrant in Hormone-Receptor-Positive (HR+), Human-Epidermal-Growth-factor-negative (HER2-) Advanced Breast Cancer Patients. The HERMIONE-7 Trial
Brief Title: Study Evaluating Abemaciclib + Aromatase Inhibitors in HR+, HER2- Advanced Breast Cancer Patients (HERMIONE-7)
Acronym: HERMIONE-7
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in patient recruitment
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERMIONE-7
Record Dates: First submitted 2019-12-17; First posted 2020-01-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer
Keywords: abemaciclib; Hormone-Receptor-Positive (HR+); Human-Epidermal-Growth-factor-negative (HER2-)
MeSH Terms: interventions — abemaciclib; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abemaciclib + aromatase inhibitors (Experimental): Abemaciclib will be administered at 150 mg twice daily orally + Letrozole 2,5 mg daily or Anastrozole 1 mg daily
  Interventions: Drug: Abemaciclib; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib will be administered orally at 150 mg twice daily
Drug: Aromatase Inhibitors — Letrozole 2,5 mg daily or Anastrozole 1 mg daily

SUMMARY:
The HERMIONE-7 trial is a phase II, single-arm, open-label, multicenter study in HR+, HER2- advanced breast cancer patients who have received HD-FUL as first-line endocrine treatment for their metastatic disease. Patients will receive aromatase inhibitors plus Abemaciclib.

DETAILED DESCRIPTION:
Hormone receptor positive tumors represent the most common form of breast cancer and account for most of the deaths from the disease. Endocrine therapy (ET) represents the main initial therapeutic strategy for these patients and has been associated with significant clinical benefits in the majority of them.

Key-Topics for rationale:

* Fulvestrant, an Estrogen-Receptor (ER) antagonist with no known agonist effects, suppresses estrogen signaling by binding to and degrading the ER. Fulvestrant was approved as a monthly 250 mg dosing regimen based on TTP data demonstrating non-inferiority versus anastrozole in postmenopausal women whose advanced breast cancer had progressed during prior anti-estrogen therapy.
* The international CONFIRM trial compared Fulvestrant 500 mg (High-Dose Fulvestrant HD-FUL: Fulvestrant 500 mg every month with an additional 500 mg loading dose on Day 14 of the first month) with the monthly 250 mg dose and demonstrated that HD-FUL mg was associated with improved progression-free survival (PFS) and overall survival (OS) in postmenopausal women with ER-positive (ER+) advanced breast cancer whose disease had recurred or progressed after prior endocrine therapy.
* The FALCON study evaluated the efficacy and safety of HD-FUL in comparison to anastrozole in HR+, HER2- recurrent or metastatic breast cancer (MBC) patients. Median duration of PFS with HD-FUL was 16·6 months (95% CI 13·83-20·99) in the whole population and 22.3 months (95% CI 16·62-32·79) in the non-visceral one. Grade 3 or worse adverse events were reported by 51 (22%) of 228 patients receiving HD-FUL.
* Palbociclib, Abemaciclib and Ribociclib + Fulvestrant are superior to Fulvestrant alone in terms of PFS (PALOMA-3: 9.5 vs 4.6 months; MONARCH-2: 16.4 vs 9.3; MONALEESA-3: 20.5 vs 12.8) in patients who have received prior endocrine therapy for advanced disease or have relapsed during or within 1 month from adjuvant therapy.
* A descriptive study analyzed European treatment patterns for HR-positive MBC patients in real-world clinical practice in the years 2004 - 2013 showed that Fulvestrant was the initial therapy for advanced disease in 0.8 - 2.6% of the patients. However, the ongoing real-world GIM-13 AMBRA study showed that in Italy this percentage has grown up to 30%.

At the moment, no data are available regarding the activity of CDK 4/6 inhibitors in patients treated with HD-FUL as 1st-line therapy, nor are there ongoing trials in this setting.

The aim of this study is to describe the activity of Abemaciclib + aromatase inhibitors (AIs - letrozole or anastrozole) in HD-FUL pre-treated MBC patients in terms of Clinical Benefit Rate (CBR).

This is a phase II, single-arm, open-label, multicenter study in HR+, HER2- advanced breast cancer patients who have received HD-FUL as first-line endocrine treatment for their metastatic disease. Patients will receive aromatase inhibitors plus Abemaciclib.. Abemaciclib will be administered orally at 150 mg twice daily until evidence of disease recurrence or other discontinuation criteria are met, whichever occurs first, together with AIs, as per specific product instructions. The Simon's optimal two-stage design will be used for the conduction of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years of age regardless of menopausal status, who have relapsed while on prior first-line therapy with HD-FUL
2. Patients with advanced (loco-regionally recurrent, or metastatic) breast cancer not amenable to curative therapy.
3. Patient has a histological and/or cytological confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory.
4. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
5. WHO performance status of 0-2
6. Measurable disease (according to Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1) or at least one lytic bone lesion
7. The patient is able to swallow oral medications.
8. The patient has adequate organ function
9. Patient has signed ICF (ICF) obtained before any trial-related activities Patients must be able to communicate with the investigator and comply with the requirements of the study procedures.

Exclusion Criteria:

1. Patient has a known hypersensitivity to any of the excipients of Abemaciclib or letrozole/anastrozole
2. Patient who received any CDK4/6 inhibitor
3. Patient who received > 1 prior systemic hormonal therapy for advanced breast cancer; the only admitted previous therapy as 1st-line treatment is HD FUL. Note: Patients who received ≤ 28 days of letrozole or anastrozole for advanced disease prior to inclusion in this trial are eligible.
4. Patient who has not had resolution of all acute toxic effects of prior anti-cancer therapy to NCI CTCAE version 4.03 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion)
5. Patient who has received extended-field radiotherapy ≤ 4 weeks or limited field radiotherapy for palliation ≤ 2 weeks prior to start of treatment, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the patient at the investigator's discretion).
6. Patients from whom ≥ 25% (Ellis RE 1961) of the bone marrow has been previously irradiated are also excluded.
7. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of treated, basal or squamous cell carcinoma, non melanomatous skin cancer or curatively resected cervical cancer.
8. Patient with central nervous system (CNS) metastases unless they meet ALL of the following criteria:

   1. At least 4 weeks from prior therapy for CNS disease completion (including radiation and/or surgery) to starting the study treatment
   2. Clinically stable CNS lesions at the time of study treatment initiation and not receiving steroids and/or enzyme-inducing anti-epileptic medications for the management of brain metastases for at least 2 weeks
9. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection, or preexisting Crohn's disease or ulcerative colitis, or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)
10. Patient has a known history of HIV infection (testing not mandatory)
11. The patient has serious preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (such as severe renal impairment, [for example, estimated creatinine clearance <30 mL/min], interstitial lung disease, sever dyspnea at rest or requiring oxygen therapy
12. The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Exception: patients with controlled atrial fibrillation for >30 days prior to randomization are eligible. Any patient with a history of VTE (for example, DVT of the leg or arm and/or PE) will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) in HD-FUL pre-treated MBC patients treated with Abemaciclib + aromatase inhibitors (letrozole or anastrozole) | At 6 months from treatment initiation
  CBR is defined as the proportion of patients in Complete Response (CR), Partial Response (PR) or with Stable Disease (SD) >= 24 weeks (as defined by RECIST 1.1 Criteria) evaluated at 6 months from treatment initiation.

SECONDARY OUTCOMES:
Time To Progression (TTP) | Through study completion, an average of 42 months
  TTP is defined as the time from date of start of treatment to the date of event, i.e. the first documented progression or death due to underlying cancer
Overall Response Rate (ORR) | Through study completion, an average of 42 months
  ORR is defined as the proportion of patients with best overall response of CR or PR) according to RECIST 1.1.
Duration of Overall Response (DoOR) | Through study completion, an average of 42 months
  DoOR is defined as the time of initial response until documented tumor progression
Duration of Clinical Benefit (DoCB) | Through study completion, an average of 42 months
  DoCB is defined as the time of initial CB until documented tumor progression
To assess the safety profile of Abemaciclib in association with aromatase inhibitors (letrozole or anastrozole) | Through study completion, an average of 42 months
  The Medical Dictionary for Regulatory Activities (MedDRA) Version 19.0 (or higher) will be used when reporting AEs by MedDRA terms. The MedDRA Lower Level Term will be used in the treatment-emergent computation. Treatment-emergent adverse events will be summarized by System Organ Class (SOC) and by decreasing frequency of Preferred Term within SOC.

CONTACTS AND LOCATIONS:
Locations (39):
- Italy (39):
  - AOU ospedali riuniti Ancona clinica oncologica, Ancona
  - ASL di Asti D.H. - oncologia, Asti
  - IRCCS Istituto Oncologico Giovanni Paolo II, Bari
  - Ospedale Monsignor Dimiccoli, Barletta
  - ULSS 1 Belluno Ospedale San Martino, Belluno
  - ASST degli Spedali civili, Brescia
  - ASL AL - Ospedale "Santo Spirito", Casale Monferrato
  - ASST Lariana, Como
  - ASST Cremona Istituti ospitalieri Cremona, Cremona
  - AO S. Croce e Carle Ospedale di Insegnamento, Cuneo
  - ASST Monza, Ospedale di Desio, Desio
  - ULSS1 Dolomiti - Ospedale di Feltre, Feltre
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Azienda ospedaliera S. Antonio abate, Gallarate
  - AUSL di Reggio Emilia clinica oncologica Guastalla, Guastalla
  - Azienda ospedaliera cardinale Giovanni Panico, Lecce
  - ASST Lecco, Lecco
  - AUSL Toscana Nord Ovest Livorno, Livorno
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola
  - ASST Monza, Ospedale San Gerardo, Monza
  - Istituto Oncologico Veneto IRCCS, Padua
  - Ospedale La Maddalena, Palermo
  - Policlinico universitario di Palermo - oncologia medica, Palermo
  - IRCCS Fondazione Salvatore Maugeri, Pavia
  - AUSL di Piacenza Ospedale "Guglielmo da Saliceto", Piacenza
  - Arcispedale S. Maria nuova, Reggio Emilia
  - ASST Rhodense ospedale di circolo Rho, Rho
  - AUSL Romagna ospedale di Rimini, Rimini
  - Istituto Nazionale dei tumori Regina Elena- oncologia medica A, Roma
  - Istituto Nazionale dei tumori Regina Elena- oncologia medica B, Roma
  - Humanitas research hospital, Rozzano
  - Ospedale Ruggi d'Aragona, Salerno
  - ASST Valle Olona P.O. SARONNO, Saronno
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - AOU Città della salute e della scienza - Breast Unit, Torino
  - ASL Torino presidio ospedaliero Martini, Torino
  - APSS provincia autonoma di Trento Ospedale di Trento, Trento
  - ASST Settelaghi Varese, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: No